CLINICAL TRIAL: NCT02680704
Title: Mechanical Ventilation in Severe Brain Injury: The Effect of Positive End Expiratory Pressure on Intracranial Pressure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of PI
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Valerie Banner-Goodspeed, Clinical Research Administrator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015P000089
Record Dates: First submitted 2016-02-09; First posted 2016-02-11 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Intracranial Hypertension; Critical Illness; Brain Injuries; Lung Injury; Respiratory Failure; Positive-Pressure Respiration, Intrinsic
MeSH Terms: conditions — Intracranial Hypertension; Critical Illness; Brain Injuries; Lung Injury; Respiratory Insufficiency; Positive-Pressure Respiration, Intrinsic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PEEP Titration Arm (Other): PEEP titrated mechanical ventilation
  Interventions: Other: PEEP titrated mechanical ventilation

INTERVENTIONS:
Other: PEEP titrated mechanical ventilation — Enrolled patients will receive a sequential, step-wise increase in positive end-expired pressure from 5 cmH2O to 15 cmH2O. Intracranial pressure, transpulmonary pressure, vitals, and mechanical ventilator data will be measured at each increment. PEEP will be increased by increments of 5 cmH2O. The mode of mechanical ventilation (pressure or volume control), inspiratory time and fraction of inspired oxygen (FIO2) will be determined by the critical care team caring for the patient. In the event that PEEP is set > 5 cmH2O, measurements will be obtained from that starting point and increased to a maximum of 15 cmH2O. The physiologic measurements will be obtained at regular intervals (within 5 minutes at each PEEP level) throughout the PEEP titration period.

SUMMARY:
The purpose of this study is to collect physiologic data from patients with severe brain injury who require mechanical ventilation in order to describe the impact of ventilation, specifically positive end expiratory pressure (PEEP), on intracranial pressure (ICP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe brain injury (GCS 8 or less)
* Receiving mechanical ventilation
* Receiving intracranial pressure monitoring

Exclusion Criteria:

* Esophageal varices
* Esophageal trauma
* Recent esophageal surgery
* Coagulopathy (Platelets < 80k or INR> 2 )
* Other contraindication for esophageal manometry
* Already receiving PEEP > 15 cmH2O at enrollment
* Intracranial hypertension (defined as ICP > 20 mmHg)
* Decompressive hemi-craniectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02; Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Association between PEEP and ICP | Change from baseline to 20 minutes
  Intracranial pressure will be measured and recorded using the existing intracranial pressure monitoring device placed previously as part of the patient's routine care. The association between positive end expiratory pressure and intracranial pressure will be analyzed as the primary outcome.

SECONDARY OUTCOMES:
Association between transpulmonary pressure and ICP | Change from baseline to 20 minutes
  Transpulmonary pressure will be measured and recorded using an esophageal balloon catheter placed for research purposes. The association between transpulmonary pressure change with titration of PEEP and intracranial pressure will be analyzed as a secondary outcome.
Association between PEEP and cerebral hemodynamics | Change from baseline to 20 minutes
  Cerebral hemodynamic information will be recorded and calculated. The association between positive end expiratory pressure and cerebral hemodynamics will be analyzed as a secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: M. Dustin Boone, MD, Principal Investigator — Principal Investigator
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No